CLINICAL TRIAL: NCT03287726
Title: Evaluation of the Potential Impact of Probiotics on Weight Loss Maintenance in Individuals With Obesity
Brief Title: What is the Impact of Probiotics on Weight Loss Maintenance in Individuals With Obesity?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Norwegian University of Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/1297-10
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Obesity
Keywords: Probiotics; Appetite Regulation; Gastrointestinal microbiome; Caloric Restriction; Body weight maintenance; Body composition
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotics (Experimental)
  Interventions: Dietary Supplement: probiotics
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotics — NYCOPRO, a multistrain probiotic (7 strains of Lactobacilli and Bifidobacteria) sold in the Norwegian pharmacies. 2 capsules/day (one with lunch and one with dinner). 2 text messages daily as a reminder. Follow up meeting at ObeCe (St. Olavs hospital) every month with a research nurse, for weighing, blood pressure measurement and collection of probiotics dose for the following month.
  Arms: probiotics
Dietary Supplement: placebo — Placebo 2 capsules/day (one with lunch and one with dinner). 2 text messages daily as a reminder. Follow up meeting at ObeCe (St. Olavs hospital) every month with a research nurse, for weighing, blood pressure measurement and collection of probiotics dose for the following month.
  Arms: placebo

SUMMARY:
Weight loss maintenance is the biggest challenge in obesity management, with the majority of weight-reduced individuals experiencing weight regain. The intake of probiotics has been shown to help in weight loss, but its potential in maximizing weight loss maintenance remains unknown. Therefore, the main aim of this study is to investigate the impact of probiotic consumption on weight loss maintenance. Secondary aims are to investigate if the intake of probiotics influences gut microbiota, cardio-metabolic profile, appetite and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* class I or II obesity (30 kg/m2 < BMI > 40 kg/m2)
* weight stable (<2 kg variation in weight within the last 3 months)
* not currently dieting to lose weight
* dietary intervention of 1000 kcal energy restriction for 8 weeks using a powder based low energy diet product, followed by 4 week weight stabilization phase (re-introduction of food)
* women who are either post-menopausal, taking oral contraceptives or with a normal cycle (28 ± 2 days)

Exclusion Criteria:

* consumption of probiotics 6 months before taking part in the study
* pregnant
* breast-feeding
* drug or alcohol abuse within the last two years
* currently taking medication known to affect appetite or induce weight loss
* enrolled in another obesity treatment program
* history of psychological disorders
* having had bariatric surgery
* metabolic diseases (such as hypo/hyperthyroidism and diabetes type 1 or 2)
* eating disorders
* lactose intolerance
* gastrointestinal (particularly cholelithiasis), kidney, liver, lung, cardiovascular disease
* malignancies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
body composition | 9 months
  air displacement plethysmography (BodPod, COSMED, Italy)

SECONDARY OUTCOMES:
appetite suppression | 9 months
  Online Visual Analogue Scale (VAS) for the measurement of subjective feelings of appetite (hunger, fullness, desire to eat, prospective consumption)
body composition | 9 months
  Bioelectrical impedance analysis (BIA)
resting metabolic rate | 9 months
  indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Torstein Baade Rø, phd prof, Study Chair — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Martins C, Roekenes J, Salamati S, Gower BA, Hunter GR. Metabolic adaptation is an illusion, only present when participants are in negative energy balance. Am J Clin Nutr. 2020 Nov 11;112(5):1212-1218. doi: 10.1093/ajcn/nqaa220. PMID 32844188